CLINICAL TRIAL: NCT04804410
Title: Determination of Dielectric Properties of Matched Tissue Samples From Thoracic Malignancies and Corresponding Normal Tissues
Brief Title: Dielectric Properties of Matched Tissue Samples From Thoracic Malignancies and Corresponding Normal Tissues
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: NovoCure Ltd. (Industry)
Responsible Party: Principal Investigator, Joseph S. Friedberg, MD, Head, Division of Thoracic Surgery, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00094059
Record Dates: First submitted 2021-03-02; First posted 2021-03-18 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Lung Cancer; Esophageal Cancer; Mesothelioma; Lung
Keywords: Dielectric Properties; Thoracic Malignancies
MeSH Terms: conditions — Lung Neoplasms; Esophageal Neoplasms; Mesothelioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dielectric Properties of Tissue Samples from Thoracic Malignancies and Corresponding Normal Tissues (Experimental): Our plan is to analyze 3-5 tissue probes acquired from 30 patients with a variety of thoracic malignancies. The investigators will plan to acquire tissue from each type of malignancy including: lung cancer, esophageal cancer and pleural based tumors. Tissue will be acquired in the operating room. Impedance measurements will be collected on multiple sections of excised tissue and will be translated into dielectric properties. After acquisition of data, the investigators will assess the data and continue to acquire patients to obtain significant estimates of overall tissue properties in each type of tumor. After undergoing an informed consent process in accordance with IRB approval, patients with be formally enrolled. All tumor electric property data will be stored securely and remain anonymous of patient identifying data.
  Interventions: Device: LCR Meter (Brand: Keysight, Serial Number:E498AL)

INTERVENTIONS:
Device: LCR Meter (Brand: Keysight, Serial Number:E498AL) — The LCR meter is used for electric property analysis of tissues. It works by measuring impedance on multiple sections of excised tissue and translating those measurement into dielectric properties.

SUMMARY:
The purpose of the Dielectrics Properties of Thoracic Malignancies Study (DPTMS) is to provide a wealth of knowledge for investigators involved in establishing a new and effective treatment for a variety of solid tumors using tumor treatment fields. It is intended to provide biospecimen (tumor/healthy) together with demographic data (age, sex, race, occupational history, and other epidemiologic information), and clinical data (stage, treatment, survival information, and annotated CT's). Our specific aims are to test the following hypotheses: 1) Electric properties of thoracic tumors differ from electric properties of surrounding healthy tissue 2) Different tumor types will have different electric properties 3) Electric properties of individual tumors are heterogeneous 4) Electric properties of tumors are related to the structure and composition of the underlying tissue 5) Use of standard medical imaging data (CT) will permit mapping of electric properties.

DETAILED DESCRIPTION:
Thoracic malignancies represent a significant burden of disease in the US population. Lung cancer, for example, is the most common cause of cancer mortality in the US among both men and women and long-term survival remains poor with a 5-year survival rate less than 20%. There is significant need for additional therapeutic options for all stages of patients. Esophageal cancer, although less common in the US with an incidence of 1% among new cancer diagnosis, also has significant mortality with a similar survival rate of about 20% at 5 years. There are a variety of additional thoracic malignancies that contribute to morbidity and mortality of the US population including mesothelioma and other pleural based cancers and thymoma. All of these thoracic malignancies pose unique challenges that have limited the effectiveness of current therapies, necessitating the development of new and innovative approaches.

Tumor treatment fields (TTF) have recently been established as a new and effective treatment for a variety of solid tumor malignancies. TTF provides a unique ability to deliver targeted and sustained therapy via an LCR meter. TTF has shown promise for some of the most aggressive malignancies such as glioblastoma and therefore should be considered for aggressive thoracic malignancies as well. In order to develop a TTF protocol that is both efficient and efficacious, the electric field properties of target tumors must be understood. Although well established for some tumors, the complete electric properties of thoracic malignancies as they apply to TTF is still not fully understood. The proposed project is to address this gap of knowledge.

Our plan is to analyze 3-5 tissue probes acquired from 30 patients with a variety of thoracic malignancies. Tissue will be acquired in the operating room and will be analyzed immediately. The investigators will plan to acquire tissue from each type of malignancy including: lung cancer, esophageal cancer and pleural based tumors. After acquisition of data, the investigators will assess the data and continue to acquire patients to obtain significant estimates of overall tissue properties in each type of tumor. The investigators will offer all patients at our center undergoing resection of thoracic malignancies the opportunity to participate in the study. After undergoing an informed consent process in accordance with IRB approval, patients with be formally enrolled. The LCR meter used for electric property analysis of the tissue will be positioned on and secured to a movable cart so that it can be brought to the operating room for rapid tissue analysis following surgical excision of the tumor. Impedance measurements will be collected on multiple sections of excised tissue and will be translated into dielectric properties. All tumor electric property data will be stored securely and remain anonymous of patient identifying data.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of thoracic malignancies
* Able to provide informed consent
* Scheduled for diagnostic or treatment related surgical procedure

Exclusion Criteria:

* Inability to undergo surgery
* Unable to provide informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Impedance measurements in different frequencies | During Surgery
  The impedance measurements in different frequencies will be collected on multiple sections of excised tissue and will be translated into dielectric properties. The conductivity and relative permittivity measurements in frequencies range (20Hz-1MHz) of tissues will be collected and analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Friedberg, MD, FACS, Principal Investigator — University of Maryland, Baltimore

IPD SHARING:
Plan to Share IPD: Yes
The following information will be recorded from all samples and provided to Novocure Ltd; 1) Type of tumor tissue 2) Measured electric properties 3) ID/ serial number connecting sample to annotated CT image
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Individual participant data (de-identified data) would be shared with Novocure Ltd indefinitely.
Access Criteria: All individual participant data (de-identified) would be stored on a secure database and shared with Novocure Ltd.

REFERENCES:
- [Background] Wenger C, Salvador R, Basser PJ, Miranda PC. The electric field distribution in the brain during TTFields therapy and its dependence on tissue dielectric properties and anatomy: a computational study. Phys Med Biol. 2015 Sep 21;60(18):7339-57. doi: 10.1088/0031-9155/60/18/7339. Epub 2015 Sep 9. PMID 26350296
- [Background] Gabriel C, Peyman A, Grant EH. Electrical conductivity of tissue at frequencies below 1 MHz. Phys Med Biol. 2009 Aug 21;54(16):4863-78. doi: 10.1088/0031-9155/54/16/002. Epub 2009 Jul 27. PMID 19636081
- [Background] Kirson ED, Dbaly V, Tovarys F, Vymazal J, Soustiel JF, Itzhaki A, Mordechovich D, Steinberg-Shapira S, Gurvich Z, Schneiderman R, Wasserman Y, Salzberg M, Ryffel B, Goldsher D, Dekel E, Palti Y. Alternating electric fields arrest cell proliferation in animal tumor models and human brain tumors. Proc Natl Acad Sci U S A. 2007 Jun 12;104(24):10152-7. doi: 10.1073/pnas.0702916104. Epub 2007 Jun 5. PMID 17551011
- [Background] Kirson ED, Gurvich Z, Schneiderman R, Dekel E, Itzhaki A, Wasserman Y, Schatzberger R, Palti Y. Disruption of cancer cell replication by alternating electric fields. Cancer Res. 2004 May 1;64(9):3288-95. doi: 10.1158/0008-5472.can-04-0083. PMID 15126372
- [Background] Mun EJ, Babiker HM, Weinberg U, Kirson ED, Von Hoff DD. Tumor-Treating Fields: A Fourth Modality in Cancer Treatment. Clin Cancer Res. 2018 Jan 15;24(2):266-275. doi: 10.1158/1078-0432.CCR-17-1117. Epub 2017 Aug 1. PMID 28765323
- [Background] Pless M, Droege C, von Moos R, Salzberg M, Betticher D. A phase I/II trial of Tumor Treating Fields (TTFields) therapy in combination with pemetrexed for advanced non-small cell lung cancer. Lung Cancer. 2013 Sep;81(3):445-450. doi: 10.1016/j.lungcan.2013.06.025. Epub 2013 Jul 23. PMID 23891283
- [Background] Ceresoli GL, Aerts JG, Dziadziuszko R, Ramlau R, Cedres S, van Meerbeeck JP, Mencoboni M, Planchard D, Chella A, Crino L, Krzakowski M, Russel J, Maconi A, Gianoncelli L, Grosso F. Tumour Treating Fields in combination with pemetrexed and cisplatin or carboplatin as first-line treatment for unresectable malignant pleural mesothelioma (STELLAR): a multicentre, single-arm phase 2 trial. Lancet Oncol. 2019 Dec;20(12):1702-1709. doi: 10.1016/S1470-2045(19)30532-7. Epub 2019 Oct 15. PMID 31628016